CLINICAL TRIAL: NCT01582880
Title: The Use of Riboflavin/Ultraviolet A Cross-linked Human Donor Corneas as Carriers for the Boston Keratoprosthesis
Brief Title: Use of Cross-linked Donor Corneas as Carriers for the Boston Keratoprosthesis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joseph B. Ciolino, MD (Other)
Responsible Party: Sponsor-Investigator, Joseph B. Ciolino, MD, Principal Investigator, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-03-020
Record Dates: First submitted 2012-04-10; First posted 2012-04-23 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Chemical Injuries; Unspecified Complication of Corneal Transplant; Autoimmune Diseases; Ocular Cicatricial Pemphigoid; Stevens Johnson Syndrome; Lupus Erythematosus, Systemic; Rheumatoid Arthritis; Other Autoimmune Diseases
Keywords: Keratoprosthesis; sterile cornea ulcer
MeSH Terms: conditions — Autoimmune Diseases; Pemphigoid, Benign Mucous Membrane; Stevens-Johnson Syndrome; Lupus Erythematosus, Systemic; Arthritis, Rheumatoid | interventions — Riboflavin; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Riboflavin Cross-linked donor cornea (Experimental): the donor cornea used as a carrier for the Boston Keratoprosthesis will undergo crosslinking treatment before being trephined and prepared for implantation with the Keratoprosthesis.
  Interventions: Drug: Riboflavin

INTERVENTIONS:
Drug: Riboflavin — Used to treat donor cornea before implantation
  Other Names: Riboflavin (vitamin B2) 0.1% solution

SUMMARY:
The purpose of the pilot study is to test the efficacy and safety of riboflavin/Ultraviolet A (UVA) cross-linked human donor corneas as carriers for the Boston Keratoprosthesis (Boston KPro) in patients with higher risk for corneal melting (keratolysis).

DETAILED DESCRIPTION:
The corneal cross-linking technique has been shown to strengthen the cornea and resist degradation by the body's own enzymes. The use of highly-resistant donor corneas is meant to eliminate the serious post-operative complication of corneal melting (keratolysis) that repeatedly occurs in Boston KPro patients with severe ocular burns, autoimmune and cicatrizing diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent and comply with study assessments for the full duration of the study.
2. Age > 18 years.
3. A negative urine pregnancy test.
4. Candidate for a Boston Keratoprosthesis/Corneal transplant.
5. Generally good stable overall health.
6. Patients with an eye at risk for a cornea sterile ulcer which includes:

   * Chemical injuries.
   * Autoimmune diseases (ocular cicatricial pemphigoid, Stevens Johnson Syndrome, systemic lupus erythematosus, rheumatoid arthritis, or other autoimmune diseases).
   * History of previous sterile corneal ulceration requiring a cornea transplant.

Exclusion Criteria:

1. Age < 18 years.
2. Inability to provide written informed consent and comply with study assessments for the full duration of the study.
3. Pregnant or lactating women.
4. No or minimal tear production.
5. Ocular or periocular malignancy.
6. Inability to wear a contact lens due to lid abnormalities or shortened fornix.
7. Signs of current infection, including fever and current treatment with antibiotics.
8. Participation in another simultaneous medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ciolino, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Riboflavin Cross-linked Donor Cornea
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Riboflavin Cross-linked Donor Cornea
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (NA) — Standard Deviation is not applicable for a single participant
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
corneal thickness measured at 1mm one day post op [Number; unit: µm] — "corneal thickness measured at 1mm one day post op" is the baseline measurement for this study. This study evaluated cross-linked cornea tissue versus standard of care cornea tissue after transplant procedure. Therefore the measurement at one day post op is the baseline measurement.
  µm | 730
corneal thickness measured at 2mm one day post op [Number; unit: µm] — "corneal thickness measured at 2mm one day post op" is the baseline measurement for this study. This study evaluated cross-linked cornea tissue versus standard of care cornea tissue after transplant procedure. Therefore the measurement at one day post op is the baseline measurement.
  µm | 940

OUTCOME MEASURES:

1. Primary Outcome: Changes in Corneal Thickness at 1 Millimeter
Description: The average carrier graft thickness over the first year of postoperative follow-up. The corneal thickness was measured at each visit using AS-OCT imaging 1 mm away from the KPro stem at 3, 6, 9, and 12 o'clock. The individual corneal thickness measurements (3, 6, 9, and 12 o'clock) where then averaged. The average corneal thickness measurements for week 4, 6, 26, 32 and 52 are reported below.
Time Frame: measured at week 4, 6, 26, 32, 52
Population: 52 year old white male patient
Measure: Number; unit: micrometer
Groups:
- Riboflavin Cross-linked Donor Cornea: The donor cornea used as a carrier for the Boston Keratoprosthesis underwent crosslinking treatment before being trephined and prepared for implantation with the Keratoprosthesis.
  Riboflavin: Used to treat donor cornea before implantation
Arm/Group | Riboflavin Cross-linked Donor Cornea
Number analyzed (Participants) | 1
micrometer
  week 4 corneal thickness | 730
  week 6 corneal thickness | 760
  week 26 corneal thickness | 700
  week 32 corneal thickness | 720
  week 52 corneal thickness | 680

2. Primary Outcome: Changes in Corneal Thickness at 2 Millimeter
Description: The average carrier graft thickness over the first year of postoperative follow-up. The corneal thickness was measured at each visit using AS-OCT imaging 2 mm away from the KPro stem at 3, 6, 9, and 12 o'clock. The individual corneal thickness measurements (3, 6, 9, and 12 o'clock) where then averaged. The average corneal thickness measurements for week 4, 6, 26, 32 and 52 are reported below.
Time Frame: measured at week 4, 6, 26, 32, 52
Population: 52 year old white male patient
Measure: Number; unit: micrometer
Arm/Group | Riboflavin Cross-linked Donor Cornea
Number analyzed (Participants) | 1
micrometer
  week 4 corneal thickness | 940
  week 6 corneal thickness | 860
  week 26 corneal thickness | 820
  week 32 corneal thickness | 795
  week 52 corneal thickness | 780

3. Secondary Outcome: Number of Occurrences of Vitritis (Sterile or Infectious) Ulcers
Description: Number of occurrence of vitritis (sterile or infectious) ulcers. Incidences of ulcers were collected by way of slit lamp photography from time of surgery to final visit.
Time Frame: post op week 52
Population: 52 year old white male
Measure: Number; unit: occurrences
Arm/Group | Riboflavin Cross-linked Donor Cornea
Number analyzed (Participants) | 1
occurrences | 0

4. Secondary Outcome: Ocular Safety
Description: Incidence and severity of ocular adverse events during the study (ophthalmic examination, adverse events spontaneously reported)
Time Frame: measured at day 1, and week 1, 4, 8, 12, 16, 24, 36, 52
Population: 52 year old white male
Measure: Number; unit: Incidences
Arm/Group | Riboflavin Cross-linked Donor Cornea
Number analyzed (Participants) | 1
Incidences | 0

5. Secondary Outcome: Systemic Safety
Description: Incidence and severity of systemic adverse events during the study (clinical laboratory, adverse events spontaneously reported).
Time Frame: measured at day 1, and week 1, 4, 8, 12, 16, 24, 36, 52
Population: 52 year old white male
Measure: Number; unit: Incidences
Arm/Group | Riboflavin Cross-linked Donor Cornea
Number analyzed (Participants) | 1
Incidences | 0

ADVERSE EVENTS:
Time Frame: This study enrolled one study subject. The study subject was followed for Adverse Events from the time of signing the study informed consent form 2/12/2013 to one year post surgery 3/13/2014
Arm/Group | Riboflavin Cross-linked Donor Cornea
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes